CLINICAL TRIAL: NCT05436587
Title: Identification of The Novel Mutations and A Comprehensive Analysis of The Phenotype and Genetic Etiology Underlying Unclassifiable Inherited Bone Marrow Failure Syndromes With Bone Fragility Fractures
Brief Title: Mutations and Phenotypes of Unclassifiable Inherited Bone Marrow Failure Syndromes
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Collaborators: Kyoto University (Other); Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ibrahim Yousef, Principal Investigator, Sohag University
Other Study IDs: Soh-Med-22-01-40
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Inherited BMF Syndrome
MeSH Terms: conditions — Congenital Bone Marrow Failure Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: The whole-exome sequencing — Exome sequencing will be performed at the Division of Hematopoietic Disease Control, The Institute of Medical Science, The University of Tokyo, Tokyo, Japan and will be analyzed at Institute for the Advanced Study of Human Biology (WPI-ASHBi), Kyoto University, Japan.
  Other Names: Radiologic assessment; Histopathological studies of BM biopsies; • Chromosomal fragility testing

SUMMARY:
Inherited bone marrow failure syndromes (IBMFSs) are a diverse collection of genetic illnesses characterized by various degrees of peripheral cytopenias due to defective single-lineage or multi-lineage hematopoiesis, it can manifest itself at birth or later in life.

DETAILED DESCRIPTION:
Studying the genetic etiology underlying unclassifiable IBMFSs with bone fragility fractures should be useful for clarifying the undiagnosed pathophysiological mechanisms and other accessory factors to improve the diagnosis, follow-up, prognosis, and management of these patients as well as prevent future complications.

Moreover, early diagnosis of risk factors of unusual presentations of IBMFSs will be a useful tool for better treatment strategy.

In addition, along with typical IBMFSs, novel clinical entities must be included in an overall molecular portrait of IBMF disorders. As a result, comprehensive genetic analysis will be effective in establishing an accurate genetic diagnosis at medical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed a two-generational family with IBMFSs presented with signs and symptoms of bone fragility fractures and admitted or treated in Hematology Division at Internal Medicine Departments of various university hospitals will be screened for enrollment in this study.
* The investigators will invite the entire family for testing for IBMFSs mutations, and three additional family members consented to participate in this study.

Exclusion Criteria:

* • Patients will be diagnosed with paroxysmal nocturnal hemoglobinuria

  * Patients will be diagnosed with de novo myelodysplastic syndrome
  * IBMFSs-patients will refuse to consent to this study.
  * Serologic evidence of recent virus infection as hepatitis A (HAV), HBV, HCV, HEV, cytomegalovirus (CMV), Epstein-Barr virus (EBV), or positive test for HIV.
  * IBMFSs patients with severe systemic diseases (such as cardiovascular, renal, and hepatic disease) or surgical/medical conditions that might interfere with follow-up instructions.
  * IBMFs patients with psychiatric disorders or a history of drug abuse,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The candidate patients who will have evidence of unclassifiable IBMFSs and/or will present with manifestations suggesting IBMFSs and agree to comply with follow-up instructions will be screened for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Progression of pancytopenia | Two year after diagnosis
  Progression of pancytopenia severity
Number of Participants with Fragility Fractures | Two year after diagnosis
  occurrence of the Fragility Fractures
Number of Participants with Malignancy transformation | Two year after diagnosis
  Occurrence of hematological or solid malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud I Yousef, PhD, Principal Investigator — Faculty of Medicine, Sohag University
Locations (1):
- , Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sieff CA. Acquired and Inherited Bone Marrow Failure Syndromes. Hematol Oncol Clin North Am. 2018 Aug;32(4):xiii-xiv. doi: 10.1016/j.hoc.2018.05.001. No abstract available. PMID 30047424
- [Derived] Elbadry MI, Tawfeek A, Hirano T, El-Mokhtar MA, Kenawey M, Helmy AM, Ogawa S, Mughal MZ, Nannya Y. A rare homozygous variant in TERT gene causing variable bone marrow failure, fragility fractures, rib anomalies and extremely short telomere lengths with high serum IgE. Br J Haematol. 2024 Mar;204(3):1086-1095. doi: 10.1111/bjh.19176. Epub 2023 Nov 5. PMID 37926112